CLINICAL TRIAL: NCT03715478
Title: A Phase 1/2 Multi-Center, Open Label, Dose Escalation Study to Determine the RP2D, Safety and Efficacy of GSK2857916 in Combination With Pomalidomide and Low-Dose Dexamethasone in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Multi-Center Study of GSK2857916 in Combination With Pomalidomide and Dex
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canadian Myeloma Research Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMRG 007; ALGONQUIN (Other: CMRG)
Record Dates: First submitted 2018-10-02; First posted 2018-10-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — belantamab mafodotin; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSK2857916 with Pomalidomide and Dexamethasone (Experimental): This will be a single arm study of GSK2857916 administered with pomalidomide and dexamethasone. GSK2857916 will be administered intravenously either on Day 1 of each 28 day cycle (Single Dose) or on Days 1 and 8 (Split Dose) and up to 4 dose levels will be evaluated during the phase I portion. Pomalidomide will be administered orally on Days 1-21 at 4 mg. Dexamethasone will be administered orally at 40 mg for patients ≤ 75 years old or 20 mg for patients older than 75 on days 1, 8, 15, 22.
  Interventions: Drug: GSK2857916 with Pomalidomide and Dexamethasone

INTERVENTIONS:
Drug: GSK2857916 with Pomalidomide and Dexamethasone — Recommended phase 2 dose (RP2D) of GSK2857916 determined by the phase 1 portion of study will be administered in combination with pomalidomide (approved dose and schedule) and dexamethasone until progression of disease.
  Other Names: Pomalyst

SUMMARY:
This is a Phase 1/2, multi-centre, single-arm, open-label, dose-escalation study that will evaluate the safety and efficacy of IV GSK2857916 in combination with PO pomalidomide and low-dose PO dexamethasone in subjects with relapsed and/or refractory MM.

DETAILED DESCRIPTION:
This is a Phase 1/2, multi-centre, single-arm, open-label, dose-escalation study that will evaluate the safety and efficacy of IV GSK2857916 in combination with PO pomalidomide and low-dose PO dexamethasone in subjects with relapsed and/or refractory MM.

This study will consist of a Part 1 dose-finding portion and a Part 2 expansion phase. Part 1 will determine the starting dose and schedule to be used in Part 2. All subjects will receive GSK2857916 given IV either on Day 1 (Single Dose) or on Days 1 and 8 (Split Dose) in combination with pomalidomide and dexamethasone administered orally in 28-day treatment cycles. Treatment will be administered as long as there is clinical benefit.

The Part 1 portion of the study will determine the MTD and/or RP2D and dose limiting toxicities (DLTs) of GSK2857916 administered in combination with pomalidomide and dexamethasone. The following dose levels of GSK2857916 in combination with 4 mg of pomalidomide and low-dose dexamethasone are to be tested in this study: 2.5 mg/kg either Single Dose (dose level 1a) or Split Dose (dose level 1b), 1.92 mg/kg Single Dose (dose level -1), and 3.4 mg/kg Split Dose (dose level 2). The Part 1 segment of the study will follow a standard 3 + 3 dose escalation design and will include assessment of the safety of treatment between each dose cohort by the Safety Review Committee (SRC) consisting of the Study Investigators and the Sponsor.

When the SRC has determined the RP2D of GSK2857916, the Part 2 portion of the study will be initiated. Pomalidomide will be administered based on the current approved dose and schedule: 4 mg PO QD on Days 1 to 21 of a 28-day cycle. The starting dose of dexamethasone will be 40 mg QD on Days 1, 8, 15 and 22 of each 28-day cycle for subjects who are ≤ 75 years of age. For Subjects who are > 75 years of age, the starting dose of dexamethasone is 20 mg QD on Days 1, 8, 15, and 22. GSK2857916 will be administered at the RP2D and treatment will continue until progressive disease (PD) or toxicity requiring discontinuation of study drug. Efficacy assessments will be conducted every cycle for the duration of the treatment period. After discontinuation from treatment, follow up will continue by phone or in person until progression from the next line of treatment or death to a maximum of 36 months after enrolment for determination of PFS2 and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form (ICF).
2. Must be ≥ 18 years of age at the time of signing the ICF.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Documented diagnosis of MM and relapsed and/or refractory disease with:

   * Have undergone stem cell transplant, or have been considered transplant ineligible
   * Previously treated with two or more prior lines of treatment that must have included lenalidomide and a proteasome inhibitor (in separate regimens or in combination). Induction therapy followed by ASCT and consolidation/maintenance will be considered as one line.
   * Documented evidence of progressive disease (PD) after achieving at least stable disease (SD) for ≥ 1 cycle during a previous MM treatment (i.e., relapsed MM) and/or
   * Disease progression during or within 60 days from the end of the most recent MM treatment (i.e., refractory MM).
5. Subjects with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met:

   * transplant was > 100 days prior to study enrolment
   * no active infection
6. Subjects with measurable disease defined as at least one of the following (these baseline laboratory studies for determining eligibility must be obtained within 28 days prior to start of study drug):

   * Serum M-protein ≥ 5 g/l
   * Urine M-protein ≥ 200 mg/24 h
   * Serum free light chains (FLC) assay: Involved FLC level ≥ 100 mg/l and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
7. Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
8. Females of child-bearing potential (FCBP) must have two negative serum pregnancy test, as described in Appendix 1 for the RevAid® program. FCBP and males must either commit to continued abstinence from heterosexual intercourse or must abide by birth control requirements 120 days post discontinuation of treatment as described in Appendix 1 for the RevAid® program.
9. Men with a female partner and females of childbearing potential must agree to use effective contraception as described in Appendix 1 from the time of first dose of study until 120 days (females) and 140 days after the last dose of study treatment to allow for clearance of any altered sperm.
10. Must be able to take acetylsalicylic acid (ASA) (81 or 325 mg) daily as prophylactic anticoagulation. Subjects intolerant to ASA may use low molecular weight heparin or alternative anticoagulant.
11. Must be registered into the mandatory RevAid® program and be willing and able to comply with the requirements of the RevAid® program.
12. Able to take oral medications.
13. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be ≤Grade 1 at the time of enrollment except for alopecia or be deemed to be irreversible (for example, steroid induced cataracts).
14. The following laboratory results must be met within 10 days of first study drug administration:

    * Absolute neutrophil count (ANC) > 1.0 x 109/L. G-CSF cannot be given within 10 days prior to screening.
    * Serum ALT ≤ 2.5 x upper limits of normal (ULN).
    * eGFR (MDRD) ≥ 40 mL/min (Appendix 2).
    * Platelet count > 75 x 109/L. Platelet transfusions to help subjects meet eligibility criteria are not allowed within 10 days before study enrolment.
    * Hemoglobin ≥ 80 g/L.
    * Total bilirubin ≤ 1.5 x ULN, unless known to have Gilbert's disease. If Gilberts, isolated bilirubin > 1.5 and < 3xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
    * Albumin/creatinine ratios (spot urine) <500mg/g (56 mg/mmol)
    * Albumin ≥ 20 g/L.

Exclusion Criteria:

1. Prior pomalidomide or BCMA therapy use.
2. History of allegeneic transplant
3. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
4. Pregnant or lactating females.
5. Subjects with previous or concurrent malignancies are allowed only if the second tumor is not contributing to the subject's illness. The subject must not be receiving active therapy, other than hormonal therapy for this disease and the disease must be considered medically stable for at least 2 years.
6. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect subject's safety). Subjects with isolated proteinuria resulting from MM are eligible, provided they fulfil criteria given in inclusion criteria (i.e. albumin/creatinine < 500 mg/ g (56 mg/mmol).
7. Evidence of cardiovascular risk including any of the following:

   1. QTc interval ≥ 470 msecs. NOTE: The QT interval should be corrected for the heart rate by Fridericia's formula (QTcF)
   2. Evidence of current clinically significant uncontrolled arrhythmias; including clinically significant ECG abnormalities; including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
   3. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening.
   4. Class III or IV heart failure as defined by the New York Heart Association functional classification system (Appendix 3)
   5. Uncontrolled hypertension
8. Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at screening or within 3 months prior to first dose of study treatment. Participants with positive hepatitis B core antibody (HBcAb) can be enrolled, only if confirmatory negative Hepatitis B DNA is obtained AND patient is on hepatitis B prophylaxis (tenofovir or entecavir) before first dose of study drug.
9. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment. Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
10. Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria.
11. Current corneal epithelial disease except for mild punctate keratopathy (mild punctate keratopathy is allowed).
12. Known active infection requiring antibiotic, anti-viral or anti-fungal treatment.
13. Evidence of active mucosal or internal bleeding.
14. Hypersensitivity to thalidomide, lenalidomide (such as Steven Johnson Syndrome) or intolerance to dexamethasone. Hypersensitivity, such as rash, that can be medically managed is allowable.
15. Peripheral neuropathy ≥ Grade 2 despite supportive therapy.
16. Radiotherapy (with the exception of local, palliative radiotherapy for management of pain) or systemic therapy (standard or biologic anticancer agent) within 14 days of initiation of study drug treatment.
17. Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drug.
18. Any major surgery within the last 4 weeks.
19. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2857916 or any of the components of the study treatment.
20. Intolerance to prednisone or dexamethasone that would preclude the patient from taking the full starting dose of dexamethasone as described in the protocol (Section 6.2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 9 months
  RP2D and schedule of GSK2857916 for Part 2 will be determined by Part 1 of the study
Overall Response Rate (ORR) | 60 months
  Overall response rate will be the percentage of patients achieving partial response or better according to IMWG response criteria

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | 60 months
  Treatment Emergent Adverse Events occurring during the study will be evaluated according to CTCAE version 5.0 to determine the safety of the study treatment
Progression Free Survival | 60 months
  Progression Free Survival according to IMWG criteria will be evaluated
Maximum tolerated dose (MTD) | 9 months
  Adverse Events occurring during the first cycle of study treatment will be evaluated against a predefined dose limiting toxicities to determine the maximally tolerated dose (MTD)

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trudel S, McCurdy A, Louzada ML, Parkin S, White D, Chu MP, Kotb R, Mian H, Othman I, Su J, Khan A, Gul E, Reece D. Belantamab mafodotin, pomalidomide and dexamethasone in refractory multiple myeloma: a phase 1/2 trial. Nat Med. 2024 Feb;30(2):543-551. doi: 10.1038/s41591-023-02703-y. Epub 2024 Jan 4. PMID 38177852